CLINICAL TRIAL: NCT05089175
Title: The Investigation of the Prediction Model and Prevention Strategy of Serious Pregnancy Complications in Hypertensive Disorders of Pregnancy Based on the Chinese Population
Acronym: HDP-RPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: ChiCTR2100048266
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Hypertensive Disorder of Pregnancy; Pregnancy Complications
Keywords: Risk prediction; Preeclampsia Prevention; Hypertensive disorders of pregnancy
MeSH Terms: conditions — Toxemia; Pregnancy Complications | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 29 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women at high risk for preeclampsia: Using FIGO recommended preeclampsia screening model for the first-trimester which combined maternal risk factors, mean arterial pressure, placental growth factor, uterine artery pulsatility index to evaluate pregnant's risk for preeclampsia. Risk value≥1/100 is defined as screened high risk.
  Interventions: Drug: Low-dose aspirin
- Women at low risk for preeclampsia: Using FIGO recommended preeclampsia screening model for the first-trimester which combined maternal risk factors, mean arterial pressure, placental growth factor, uterine artery pulsatility index to evaluate pregnant's risk for preeclampsia. Risk value<1/100 is defined as screened low risk.

INTERVENTIONS:
Drug: Low-dose aspirin — FIGO adopts and supports that in high-risk women, defined by the first-trimester combined test, aspirin ~150 mg/night should be commenced at 11-14+6 weeks of gestation until either 36 weeks of gestation, when delivery occurs, or when pre-eclampsia is diagnosed.
  Groups: Women at high risk for preeclampsia

SUMMARY:
1. Evaluation of the efficacy of aspirin in preventing preeclampsia and its serious complications during pregnancy and postpartum. 2. To establish a risk prediction model for severe pregnancy complications in pregnant women with hypertensive disorders of pregnancy.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy (HDP) is the second leading cause of maternal death in clinical practice. The prediction and prevention of HDP and its serious complications could be a breakthrough to further reduce the maternal mortality rate in China. Aspirin (ASP) is widely used clinically as a first-line prevention program for preeclampsia (PE). However, how to determine the effectiveness of ASP prevention before the onset of PE high-risk pregnant women and adjust the risk monitoring plan accordingly has become a clinical difficult point. Two prospective and observational researches will be lauched in this study. In the first part of this study, ASP resistance test and HDP-related biomarkers will be combined to evaluate the effect of ASP on the prevention of PE from multiple dimensions, and placental pathology will be analyzed to assist evaluate, in order to more comprehensively evaluate the preventive effect of aspirin in high-risk of PE pregnant women in the first and second trimester. In the second part of this study, we aim to reduce the incidence of serious HDP complications and improve maternal and child outcomes for pregnant women with HDP who have missed HDP prediction and prevention opportunities in the first trimester, or aspirin prevention is ineffective. It is planned to establish a risk prediction model for severe pregnancy complications in pregnant women with HDP by adding other biological and physical indicators on the basis of maternal factors, in order to more accurately predict one or several severe complications of HDP over a period of time.

ELIGIBILITY:
Inclusion Criteria:Part I: Evaluation of the efficacy of aspirin in preventing preeclampsia and severe pregnancy complications 1.11-13 + 6 gestational weeks; 2.≥18 years old; 3. Monocyesis, fetal survival; 4. Agree to participate and sign the informed consent. Part II: The establishment of a risk prediction model for severe pregnancy complications of hypertensive disorders of pregnancy 1.20-36 + 6 gestational weeks 2. Diagnosed ≥1 of the following diseases ① Hypertension during pregnancy ② Preeclampsia ③ Pregnancy complicated with chronic hypertension ④ Chronic hypertension with preeclampsia 3.≥18 years old; 4. Monocyesis, fetal survival; 5. Agree to participate and sign the informed consent.

-

Exclusion Criteria:Part I: Evaluation of the efficacy of aspirin in preventing preeclampsia and severe pregnancy complications 1. Twin or multiple pregnancies; 2. Severe fetal malformation/abnormality; 3. Routine aspirin use before enrollment; 4. Have a history of aspirin contraindications, such as salicylic acid allergy, ulcerative disease of the digestive tract, and bleeding, liver cirrhosis, kidney failure, platelet count < 50 x 109 / L, hematocrit < 10%, hemophilia, congenital platelet disease, fibrinogen defects, or shortage, taking other antiplatelet agents except for aspirin, the use of anti-inflammatory drugs or the use of warfarin. 5. Patients who have been diagnosed with hypertensive disorders of pregnancy; 6. Severe mental disorder and inability to express will; 7. If she has obvious other abnormal physical signs, laboratory tests, and other clinical diseases, she is not suitable to participate in the study as judged by the researcher; 8. According to the researcher's judgment, childbirth information could not be obtained through observation and follow-up. Part II: The establishment of a risk prediction model for severe pregnancy complications of hypertensive disorders of pregnancy 1. Twin or multiple pregnancies; 2. Severe fetal malformation/abnormality; 3.Severe mental disorder and inability to express will; 4.If she has obvious other abnormal physical signs, laboratory tests, and other clinical diseases, she is not suitable to participate in the study as judged by the researcher; 5. According to the researcher's judgment, childbirth information could not be obtained through observation and follow-up.

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number diagnosed with pre-eclampsia | After 20th week of gestation
  According to the ISSHP, PE is defined as systolic blood pressure at ≥140 mm Hg and/or diastolic blood pressure at ≥90 mm Hg on at least two occasions measured 4 hours apart in previously normotensive women and is accompanied by one or more of the following new onset conditions at or after 20 weeks of gestation:
  1. Proteinuria (i.e. ≥30 mg/mol protein:creatinine ratio;
     ≥300 mg/24 hour; or ≥2 + dipstick);
  2. Evidence of other maternal organ dysfunction, including: acute kidney injury (creatinine ≥90 μmol/L; 1 mg/dL); liver involvement (elevated transaminases, e.g. alanine aminotransferase or aspartate aminotransferase >40 IU/L) with or without right upper quadrant or epigastric abdominal pain; neurological complications ; or hematological complications ; or
  3. Uteroplacental dysfunction .

SECONDARY OUTCOMES:
Number of women with adverse outcomes | After 20th week of gestation
  Maternal deaths Eclampsia ,Stroke, Parenteral infusion of third-line antihypertensive required,Myocardial infarction ,Blood oxygen saturation <90% ,Intubation required ,Pulmonary oedema ,Transfusion of blood products required,Platelet count <50× 10⁹ platelets per L,Hepatic dysfunction 1 ,Severe acute kidney injury 7 ,Dialysis required ,Placental abruption,Primary diagnosis,Pre-eclampsia ,Superimposed pre-eclampsia,Gestational hypertension,Gestational proteinuria, Small-for-gestational-age infant only,Chronic hypertension only,Chronic hypertension with a small-for-gestational-age infant,Renal disease,Transient hypertension,None of the above,Subsequent diagnosis of pre-eclampsia by adjudication team,Number with pre-eclampsia, diagnosed by adjudication,Severe pre-eclampsia,Time to diagnosis of pre-eclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Baohua Li, Phd, Study Director — Chief of obstetrics and gynecology
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poon LC, Shennan A, Hyett JA, Kapur A, Hadar E, Divakar H, McAuliffe F, da Silva Costa F, von Dadelszen P, McIntyre HD, Kihara AB, Di Renzo GC, Romero R, D'Alton M, Berghella V, Nicolaides KH, Hod M. The International Federation of Gynecology and Obstetrics (FIGO) initiative on pre-eclampsia: A pragmatic guide for first-trimester screening and prevention. Int J Gynaecol Obstet. 2019 May;145 Suppl 1(Suppl 1):1-33. doi: 10.1002/ijgo.12802. PMID 31111484
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] von Dadelszen P, Payne B, Li J, Ansermino JM, Broughton Pipkin F, Cote AM, Douglas MJ, Gruslin A, Hutcheon JA, Joseph KS, Kyle PM, Lee T, Loughna P, Menzies JM, Merialdi M, Millman AL, Moore MP, Moutquin JM, Ouellet AB, Smith GN, Walker JJ, Walley KR, Walters BN, Widmer M, Lee SK, Russell JA, Magee LA; PIERS Study Group. Prediction of adverse maternal outcomes in pre-eclampsia: development and validation of the fullPIERS model. Lancet. 2011 Jan 15;377(9761):219-27. doi: 10.1016/S0140-6736(10)61351-7. Epub 2010 Dec 23. PMID 21185591
- [Background] Navaratnam K, Alfirevic A, Jorgensen A, Alfirevic Z. Aspirin non-responsiveness in pregnant women at high-risk of pre-eclampsia. Eur J Obstet Gynecol Reprod Biol. 2018 Feb;221:144-150. doi: 10.1016/j.ejogrb.2017.12.052. Epub 2018 Jan 1. PMID 29304392